CLINICAL TRIAL: NCT01422525
Title: Effect of Trabeculectomy on Peripapillary Retinal Nerve Fiber Layer Thickness Using Spectral Domain Optical Coherence Tomography
Brief Title: Changes of the Peripapillary Retinal Nerve Fiber Layer After Filtration Surgery in Glaucoma Patients
Status: Terminated | Type: Observational
Why Stopped: short of study staff
Sponsor: University Eye Hospital, Würzburg (Other)
Responsible Party: Principal Investigator, Juliane Matlach, MD, Dr., University Eye Hospital, Würzburg
Other Study IDs: OCT-TET
Record Dates: First submitted 2011-08-21; First posted 2011-08-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Nerve Fiber Bundle Defect; Optic Nerve Diseases
MeSH Terms: conditions — Optic Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabeculectomy RNFL thickness OCT
  Interventions: Procedure: spectral domain optical coherence tomography

INTERVENTIONS:
Procedure: spectral domain optical coherence tomography — RNFL thickness measurement using spectral domain optical coherence tomography at baseline, 1, 3 and 6 months postoperatively.

SUMMARY:
At present, trabeculectomy is the most common performed and effective surgical method of filtration surgery for patients with medically uncontrolled glaucoma.

The aim of this prospective observational case study is to determine changes of the peripapillary retinal nerve fiber layer thickness using spectral domain optical coherence tomography in patients with glaucoma after surgical reduction of intraocular pressure.

DETAILED DESCRIPTION:
Baseline and postoperative measurement of the peripapillary retinal nerve fiber layer (RNFL) thickness will be performed using the following spectral domain optical coherence tomography (OCT): Cirrus™ HD-OCT (Carl Zeiss Meditec) and Spectralis® Heidelberg-Engineering.

The main outcome measures will be changes in overall and quadrant RNFL thickness with respect to reduction in intraocular pressure (IOP), correlation between RNFL thickness and alteration in visual field and predictive factors of postoperative IOP-reduction and changes of RNFL thickness.

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary open angle glaucoma
* target intraocular pressure under medical treatment was not reached
* progression of visual loss
* best corrected visual acuity of 20/100 or more
* spherical equivalent refraction of -8.0 to +4.0 D
* perimetry: less than 20% false positive answers

Exclusion Criteria:

* primary or secondary angle closure glaucoma
* congenital glaucoma
* normal tension glaucoma
* neovascular glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
change of retinal nerve fiber layer thickness | 6 months
  study was terminated

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital Wuerzburg, Würzburg, Bavaria, Germany